CLINICAL TRIAL: NCT04532411
Title: Evaluation of SARS-CoV-2 Sample Acquisition Efficiency and PPE Usage With and Without the Hexapod Personal Protective Booth
Brief Title: COVID-19 Testing Sample Acquisition Throughput and Efficiency
Acronym: HexapodBooth
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kristian R. Olson, M.D., Director, MGH Springboard Studio, Massachusetts General Hospital
Other Study IDs: QI Initiative
Record Dates: First submitted 2020-08-25; First posted 2020-08-31 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2021-02

CONDITIONS: SARS-CoV Infection; Respiratory Viral Infection; Personal Protective Equipment; Covid19
Keywords: SARS-CoV Infection; Test Sample Acquisition; Personal Protective Equipment; Personal Protective Booths; COVID19
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Booth Testing: This cohort was comprised of samples acquired as a component of outpatient SARS-CoV-2 (COVID-19) testing prior to implementation of the Hexapod personal protective booths.
- Post-Booth Testing: This cohort was comprised of samples acquired as a component of outpatient SARS-CoV-2 (COVID-19) testing after implementation of the Hexapod personal protective booths.
  Interventions: Other: Personal Protective Testing Booth

INTERVENTIONS:
Other: Personal Protective Testing Booth — Health personnel who utilize the Hexapod will remain in the booth and utilize durable gloves attached to ports through a plexiglass wall in order to administer a nasal swab for SARS-CoV-2 (COVID-19) testing. Patient escorts and housekeeping/sanitation staff perform additional tasks outside of the booth such as escorting the patient to the correct testing bay and dropping off testing vials and printed information, collect samples and deposit in the appropriate location after testing is complete, and sanitizing the patient bay before a subsequent patient is tested there.
  Other Names: Hexapod; HEPA Filtered Positive Pressure Testing Booth
  Groups: Post-Booth Testing

SUMMARY:
This QI project seeks to evaluate the relative test sample acquisition throughput, personal protective equipment utilization, and relative operational costs of provider-administered COVID-19 (SARS-CoV-2) nasal samples with and with the use of HEPA-filtered, positive pressure isolation booths.

DETAILED DESCRIPTION:
Beginning in March 2020, the MGH began outpatient testing for COVID-19 (SARS-CoV-2) utilizing a provider-administered nasal swab samples. This was administered with infection control protocols utilizing full PPE protection for health providers who would don and doff gowns and gloves with each sample acquisition. With an aim to decrease PPE usage and increase efficiency, personal protective booths with HEPA-filtered air called "Hexapods" were employed, after infection control approval, within the MGH system beginning on April 16, 2020.

Ambulatory Care Management at MGH systematically monitors testing completed and PPE usage on a weekly basis. Managers in charge of personnel changes shared necessary team structures and median salaries for different personnel involved with sample acquisition. MGH Materials management were able to report on costs related to consumable supplies used during testing.

In this investigation, this routinely collected data and averaged timed sample collection observations were used to compare before and after the Hexapod utilization.

ELIGIBILITY:
Inclusion Criteria:

* All testing performed at designated outpatient SARS-CoV-2 at Massachusetts General Hospital (MGH) testing sites beginning March 2019.

Exclusion Criteria:

* SARS-CoV-2 tests performed not performed within designated outpatient testing sites at MGH.
* Testing performed within the hospital for Emergency Department or Inpatient visits.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Outpatient SARS-CoV-2 PCR nasal swabs tests performed March through September 2020.
Sampling Method: Probability Sample
Enrollment: 28948 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Testing Throughput After Hexapod Implementation | Up to 22 weeks
  Samples acquired per hour using the Hexapod booth will be assessed as an average over a minimum of 12 weeks of testing compared to baseline throughput before April 16th.
Change in Isolation Gowns Utilized After Hexapod Utilization | Up to 22 weeks
  Gowns utilized per test will be assessed as an average over a minimum of 12 weeks of testing compared to baseline throughput before April 16th.
Change in Cost per Test After Hexapod Implementation | Up to 22 weeks
  The difference in costs of collecting test samples before and after hexapod utilization will be calculated.
Return on Investment | Up to 22 weeks
  The retail cost of the Hexapod booth will be divided by the average daily cost differential for testing observed and at maximum volume.

SECONDARY OUTCOMES:
Change in Testing Personnel Cost Per Test | Up to 22 weeks
  The difference in median shift salaries before and after Hexapod implementation will be calculated.
Change in Cost of Isolation Gowns Utilized | Up to 22 weeks
  Outcome 2 will be utilized to calculate the range of the change in cost of isolation gowns utilized compared to baseline usage for samples acquired before April 16th utilizing actual and quoted costs of gowns to Materials Management at MGH.

OTHER OUTCOMES:
Cost of Additional Consumable Supplies Utilized | Up to 22 weeks
  The Materials Management costs of durable gloves, sleeves, and filters will be be calculated from the manufacturer's recommended monthly replacements of each per booth.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no IPD collected as a part of this investigation.